CLINICAL TRIAL: NCT06721962
Title: A Phase 1/2a, Open Label, Dose Escalation Study to Evaluate the Safety and Preliminary Efficacy of TRX103 in Subjects With Moderate to Severe Treatment-Refractory Crohn's Disease
Brief Title: Treatment of Moderate to Severe Refractory Crohn's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tr1X, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRX103-02; RESTORE Study (Other: Tr1X, Inc.)
Record Dates: First submitted 2024-11-25; First posted 2024-12-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Crohns Disease
Keywords: Tr1X; RESTORE; Crohns; Crohns Disease; autoimmune; IBD; CD; chronic inflammation; gastrointestinal tract; chronic diarrhea; intestinal ulcers; abdominal pain
MeSH Terms: conditions — Crohn Disease; Abdominal Pain | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Dose level 1
  Interventions: Biological: TRX103
- Cohort 2 (Experimental): Dose level 2
  Interventions: Biological: TRX103
- Cohort 2A (Experimental): Dose level 2 with conditioning
  Interventions: Biological: TRX103; Drug: Cyclophosphamide
- Cohort 3 (Experimental): Dose level 3
  Interventions: Biological: TRX103
- Cohort 3A (Experimental): Dose level 3 with conditioning
  Interventions: Biological: TRX103; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TRX103 — TRX103 is an investigational research product that may treat and provide long term relief to individuals suffering from Crohn's Disease.
Drug: Cyclophosphamide — Low dose cyclophosphamide conditioning.
  Arms: Cohort 2A; Cohort 3A

SUMMARY:
This research study is testing an investigational research product called TRX103 as a possible treatment for individuals suffering from Crohn's Disease (CD). The primary purpose of this study is to learn how safe and effective different doses of TRX103 are when administered to individuals with CD.

DETAILED DESCRIPTION:
Please see our study website at https://www.cdclinicaltrial.com

ELIGIBILITY:
Inclusion Criteria:

1. Male and females ≥ 18 and ≤ 65 years of age at time of consent.
2. Weight of ≥ 40 kg.
3. Medical history and biological evidence of active bowel inflammation documented by:

   * Minimum of approximate 1 year of Crohn's disease diagnosis confirmed through Endoscopy, and;
   * Endoscopic evidence of CD diagnosis at least 3 months prior to and/or at Screening (SES-CD ≥ 6 for ilealcolonic or ≥ 4 isolated ileal disease by central reader)
4. Active disease defined as moderate to severe active CD at Screening defined by all of the following:

   * Evidence of mucosal inflammation, defined as SES-CD ≥ 6 (≥ 4 for subjects with isolated ileal disease), and;
   * CDAI total scores ≥ 220
5. Subject on treatment with corticosteroids may be included if they meet the following:

   * prednisone or equivalent dose ≤ 20 mg/day; or
   * budesonide ≤ 9 mg/day; or
   * has been on a stable dose for at least 7 days prior to TRX103 dose.
6. Advanced therapy-refractory disease defined by:

   Failure of two or more advanced approved therapies. Prior therapies may be inclusive of any combination of the following:
   * TNF-alpha inhibitors
   * IL-12/23 inhibitors
   * Anti-integrins
   * JAK inhibitors Failure of therapies are defined as either non-response (primary failure), complete loss of response (secondary failure) or intolerant to therapy at a dose indicated for CD.
   * Primary failure is defined as:

     * When a subject does not achieve a response after having received the induction doses of a CD approved drug per prescribing information. Induction period is defined as 12-weeks.
     * A response is defined as CDAI score that reduces by ≥ 100-point from Baseline or by Physician assessment.
   * Secondary failure, or relapse defined as:

     * Subjects who respond to the therapy or achieves remission after an induction regimen per prescribing information, but subsequently lose response or relapses during maintenance treatment.
     * Relapse is defined as an increase in the CDAI score from maintenance of ≥ 100 points and a CDAI score > 220, and/or SES-CD score ≥ 6 (or ≥ 4 if isolated ileal disease) or by Physician assessment.
   * Intolerant to therapy, defined as:

     * When a subject is unable to cope with the side effects or mechanism of actions of the treatment and/or experiences unacceptable side effects when dosed at appropriate therapeutic levels.
7. Absence of uncontrolled bacterial, viral, or fungal infection at time of enrollment.
8. Subjects must be able to understand and sign informed consent and be willing and able to complete all specified procedures and visits.

Exclusion Criteria:

1. Prior organ transplant, or allogeneic bone marrow, peripheral blood, or cord blood stem cell transplant. Note: Blood transfusion are not exclusionary if it occurred ≥ 3 years (- 3 months) of TRX103 infusion.
2. Received another investigational agent or therapy, within 28 days of planned TRX103 infusion (or 5 half-lives, whichever is longer) and/or have not recovered from treatment related toxicities.
3. Received any approved treatment for CD within the designated washout period (including off-label use of approved therapies) as per the protocol.
4. Strictures, active fistulae (including perianal), or abscess by computed tomography (CT) or magnetic resonance enterography (MRE) or Endoscopy within 6 months of Screening.
5. Positive serology for HIV.
6. Positive hepatitis-B surface antigen. Subject may be included if they are HBV PCR negative.
7. Hepatitis C virus (HCV RNA detectable in any subject with anti-HCV antibodies).
8. Subject with active or chronic recurring infections or untreated latent Tuberculosis (TB).
9. Current diagnosis of ulcerative colitis (UC), indeterminate colitis or CD isolated to colon only (the colitis must be related to CD and inclusive of ileal with or without colonic involvement).
10. Subjects with the following known complications of Crohn's Disease

    * active diverticulitis,
    * active fistulae or abscess,
    * abscess (abdominal or perianal) - abscess with no evidence of pus when pressed upon are permitted,
    * impassable fibrotic strictures - Patients with strictures passable by dilation are permitted,
    * symptomatic bowel strictures - must be confirmed via endoscopy and/or radiologically,
    * fulminant colitis,
    * toxic megacolon,
    * ostomy or ileoanal pouch - previous temporary ostomy pouch, followed by a reversal is permitted,
    * diagnosed with short gut or short bowel syndrome,
    * or any other manifestation that might require surgery while enrolled in the study.
11. Subject with surgical bowel resection within the past 3 months prior to Screening, or a history of > 2 bowel resections. Note: Surgery for temporary use of an ostomy bag or reconnection of the gut post colostomy use is not considered exclusionary, nor considered as part of the surgical resection if during the reconnection removal of tissue is required to facilitate reattachment.
12. Subjects that are pregnant, breast feeding, or aim to become pregnant during the 12 month study period. (Subjects, males and females, must agree to use a highly effective method of contraception).
13. Screening laboratory and other analyses show any of the following abnormal results:

    * Serum aspartate transaminase or alanine transaminase > 3.0 × upper limit of normal;
    * Total white blood cell count < 2,000/μL;
    * Estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula or by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation < 40 mL/min/1.73 m2;
    * Hemoglobin < 8 g/dL;
    * Bilirubin ≥ 2 x ULN;
    * Platelet count < 100,000/μL;
    * Absolute neutrophil count < 1,200/μL;
    * Absolute lymphocytes count < 750/μL.
14. Any subject with a history of significant renal, hepatic, pulmonary, or cardiac dysfunction, or on treatment to support cardiac dysfunction.
15. Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical condition or history, including laboratory results, which, in the Investigator's opinion:

    * places the subject at increased risk during participation in the study, and/or;
    * interferes with the subject's capacity to provide informed consent and their participation in the study, and/or;
    * interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of TRX103 infusion in subjects with moderate to severe treatment-refractory Crohn's Disease. | From baseline until 12 months post TRX103 infusion.
  As measured by:
  * Incidence and severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs), including CD flares (perforations, abscesses).
  * Incidence of infections, either bacterial, fungal or viral.
  * The safety of TRX103 determined by negative Replication Competent Lentivirus (RCL) at approximately 3-months, 6-months, and 12-months.

SECONDARY OUTCOMES:
Improvement in Simple Endoscopic Score for Crohn's Disease (SES-CD Score). | From baseline to Week 12 post TRX103 infusion.
  Endoscopic remission defined as:
  - Participants with ileocolonic or isolated ileal CD: SES-CD ≤ 4 points and no sub-score > 1 point in any individual variable, as scored by central reviewer at Week 12.
  OR
  - Participants with isolated ileal disease: SES-CD of 0 - 2 points, as scored by central reviewer at Week 12.
  Endoscopic response, defined as: Decrease in SES-CD ≥ 50% from Baseline at Week 12.
Improvement of CD status. | From baseline to Week 12 post TRX103 infusion.
  * Clinical remission, defined as CD Activity Index (CDAI) ≤ 150 at Week 12.
  * Clinical response, defined as ≥ 100-point reduction in CDAI score from Baseline at Week 12.
  * Proportion of subjects who discontinue corticosteroid use and achieve clinical remission at all subsequent timepoints, in subjects taking corticosteroids at Baseline.
Reduction in Fecal Calprotectin. | From baseline to Week 12 post TRX103 infusion.
  * Change from Baseline in fecal calprotectin at each timepoint.
  * Proportion of subjects with fecal calprotectin < 250 μg/mg at Week 12 or a decrease of 50% from Baseline.
Reduction of highly sensitive C-reactive protein (hs-CRP). | From baseline until 12 months post TRX103 infusion.
  Change from Baseline in hs-CRP at each timepoint.
Improvement in Patient Reported Outcomes (PRO). | From baseline until 12 months post TRX103 infusion.
  Change from Baseline in Health-Related Quality-of-Life (HRQOL) Questionnaires scores:
  * Inflammatory Bowel Disease Questionnaire (IBDQ)
  * EuroQol Group - 5 Dimension - 5 Level (EQ-5D-5L) Questionnaire
Pharmacokinetics (PK) of TRX103. | From baseline until 12 months post TRX103 infusion.
  TRX103 kinetics post infusion.
Level of Inflammation and mucosal damage | From baseline until 12 months post TRX103 infusion.
  Change from baseline in histopathological scores by Global Histologic Disease Activity Score (GHAS) and Robarts Histopathology Index (RHI).

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Northwestern, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Mount Sinai Health Systems, New York, New York
  - Cleveland Clinic, Cleveland, Ohio